CLINICAL TRIAL: NCT00595712
Title: Results of Opening-wedge High Tibial Osteotomy Using Iliac Crest Allograft Compared to Iliac Crest Autograft
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Ramin Espandar/Assistant Professor, TehranUMS
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 86-09-30-4111
Record Dates: First submitted 2008-01-05; First posted 2008-01-16 (Estimated); Last update posted 2010-05-25 (Estimated); Status verified 2010-05

CONDITIONS: Genovarum
Keywords: Genovarum; Medial opening-wedge high tibial osteotomy; allograft

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Using Iliac crest allograft in high tibial osteotomy
  Interventions: Procedure: Iliac crest allograft
- B (Active Comparator): Using iliac crest autograft in high tibial osteotomy
  Interventions: Procedure: Iliac crest autograft

INTERVENTIONS:
Procedure: Iliac crest allograft — Opening wedge osteotomy of proximal tibia with allograft from iliac crest
  Arms: A
Procedure: Iliac crest autograft — open wedge osteotomy of proximal tibia using autogenous iliac bone graft
  Arms: B

SUMMARY:
The purpose of this RCT is to determine the results of opening-wedge high tibial osteotomy in patients with genovarum deformity using iliac crest allograft compared to the results when using iliac crest autograft.

ELIGIBILITY:
Inclusion Criteria:

* Varus malalignment of knee with of without osteoarthritis: the angle between the articular surface and anatomical axis of tibia< 82 degrees
* at least 7.5 mm opening wedge is needed in medial proximal tibia to correct the deformity assessed during pre-op planning

Exclusion Criteria:

* symptomatic lateral compartment osteoarthritis of knee
* rheumatoid arthritis or other inflammatory joint diseases
* less than 100 degrees of knee range of motion
* grade III laxity in knee collateral ligaments
* history of surgery or fracture in the limb
* >15 degrees flexion contracture
* age <16 or >60 years
* >20 degrees varus deformity
* failure to attend follow-up visits
* sever bone loss in medial tibial plateau or medial femoral condyle
* >1cm joint subluxation
* presence of lateral trust during walking
* presence of patella baja
* skin derangements on medial proximal tibia
* any form of nicotine addiction

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Range of motion of the knee | before op and at follow ups
knee score (womac) | before op and at final follow up

CONTACTS AND LOCATIONS:
Overall Officials: Seyyed Mohammad J Mortazavi, M.D., Study Director — Tehran University of Medical Sciences
Locations (1):
- Imam Khomeini Hospital, Tehran, Iran

REFERENCES:
- [Derived] Haghpanah B, Kaseb MH, Espandar R, Mortazavi SMJ. No difference in union and recurrence rate between iliac crest autograft versus allograft following medial opening wedge high tibial osteotomy: a randomized controlled trial. Knee Surg Sports Traumatol Arthrosc. 2021 Oct;29(10):3375-3381. doi: 10.1007/s00167-020-06240-w. Epub 2020 Aug 24. PMID 32839849